CLINICAL TRIAL: NCT05975905
Title: A Randomized, Phase 2, Double-blind, Placebo-controlled Study to Investigate the Safety and Efficacy of KER-012 in Combination With Background Therapy in Adult Participants With Pulmonary Arterial Hypertension (TROPOS Study)
Brief Title: A Study to Investigate the Safety and Efficacy of KER-012 in Combination With Background Therapy in Adult Participants With Pulmonary Arterial Hypertension (PAH) (TROPOS Study).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Keros Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KER-012-A201
Record Dates: First submitted 2023-07-13; First posted 2023-08-04 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary arterial hypertension [PAH]
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 2:2:2:3 ratio to 1 of 4 treatment arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study in which treatment assignment will be blinded for the Investigators and any personnel (other than the unblinded pharmacist or designee) involved with the study conduct or evaluation at the investigational sites, the CRO, and the Sponsor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): KER-012 (Dose A) subcutaneously (SC) (every 4 weeks [Q4W]) Treatment Period: Dose A for 24 weeks; Extension Period: Dose A for another 72 weeks
  Interventions: Biological: Dose A KER-012
- Arm 2 (Experimental): KER-012 (Dose B) SC (Q4W) Treatment Period: Dose B for 24 weeks; Extension Period: Dose B for another 72 weeks
  Interventions: Biological: Dose B KER-012
- Arm 3 (Experimental): KER-012 (Dose C) SC (Q4W) Treatment Period: Dose C for 24 weeks; Extension Period: Dose C for another 72 weeks
  Interventions: Biological: Dose C KER-012
- Arm 4 (Placebo Comparator): Treatment Period: Placebo for 24 weeks; Extension Period: Dose B for another 72 weeks
  Interventions: Biological: Dose B KER-012; Biological: Placebo for 24 Weeks followed by Dose B KER-012 for 72 weeks

INTERVENTIONS:
Biological: Dose A KER-012 — Dose A KER-012 (Q4W);
  Arms: Arm 1
Biological: Dose B KER-012 — Dose B KER-012 (Q4W);
  Arms: Arm 2; Arm 4
Biological: Dose C KER-012 — Dose C KER-012 (Q4W);
  Arms: Arm 3
Biological: Placebo for 24 Weeks followed by Dose B KER-012 for 72 weeks — Treatment Period (24 weeks): Placebo SC (Q4W) Extension Period (72 weeks after Placebo treatment): KER-012 (Dose B) SC (Q4W)
  Arms: Arm 4

SUMMARY:
Study KER-012-A201 is Phase 2, double-blind, randomized, placebo-controlled study to determine the efficacy and safety of KER-012 compared to Placebo in adults with PAH (WHO Group 1 PH) on stable background PAH therapy. The study is divided into the Screening Period, Treatment Period, Extension Period, and Follow-Up Period.

DETAILED DESCRIPTION:
This is a randomized, phase 2, double-blind, placebo-controlled study of KER-012 in combination with background therapy in participants with PAH of World Health Organization (WHO) Group 1, functional class II-III. Participants will be randomly assigned in a 2:2:2:3 ratio to receive KER-012 (Dose A), KER-012 (Dose B), KER-012 (Dose C), or placebo by subcutaneous injection (SC) every 4 weeks for a period of 24 weeks in the placebo-controlled treatment period of the study while on background therapy. Evaluations will include changes in pulmonary vascular resistance (PVR), 6-minute walk distance (6MWD), and safety parameters. Participants who have not discontinued early from the placebo-controlled treatment period and have had their post-treatment period PVR assessment will be able to continue into the 72-week extension period in which KER-012 treated participants will continue to receive their same assigned dose level from the treatment period every 4 weeks and placebo treated participants will receive KER-012 (Dose B) every 4 weeks while on background therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants ≥ 18 years of age
* Symptomatic World Health Organization (WHO) Group 1 Pulmonary Hypertension (PH)(PAH) classified by one of the following subgroups:

  * Idiopathic pulmonary arterial hypertension (IPAH);
  * Heritable pulmonary arterial hypertension (HPAH);
  * Associated with drugs and toxins;
  * PAH associated with:

    * Connective tissue disease
    * Congenital systemic-pulmonary intracardiac shunt
* Has the following hemodynamic parameters that are consistent with the diagnosis of PAH:

  * Mean pulmonary arterial pressure (mPAP) > 20 mmHg at rest, AND
  * Pulmonary artery wedge pressure (PAWP) ≤ 15 mmHg, AND
  * PVR ≥ 5 Wood Units (400 dyn·sec·cm-5)
* Has WHO/New York Heart Association (NYHA) Functional Class (FC) II or III symptoms as assessed by the Investigator
* Must be on a stable PAH background therapy with either an endothelin-receptor antagonist (ERA) and/or a phosphodiesterase-5 inhibitor (PDE5-I) or soluble guanylate cyclase (sGC) stimulator and/or prostacyclin analogue or receptor agonist (oral/inhaled/SC/intravenous)
* 6MWD ≥ 150 and ≤ 500 meters at screening
* Provide written (signed and dated) informed consent form before the initiation of any Screening tests or procedures

Exclusion Criteria:

* Evidence or history of left ventricular dysfunction and/or clinically significant cardiac disease
* Has pulmonary function tests (PFTs) with evidence of significant obstructive or parenchymal lung disease
* Evidence of thromboembolic disease assessed by ventilation perfusion (V/Q) lung scan or other local standard of care diagnostic evaluation at the time of PAH diagnosis or after
* Has uncontrolled systemic hypertension
* Hemoglobin < 9 g/dL at Screening
* Prior heart or heart-lung transplants, active on the lung transplant list, or life expectancy of < 12 months per Investigator assessment
* Diagnosis of pulmonary veno-occlusive disease or pulmonary capillary hemangiomatosis
* Initiation or discontinuation of an exercise program for cardiopulmonary rehabilitation within 90 days prior to Baseline or planned initiation during the study
* Prior participation in a KER-012 study or prior treatment with a therapy targeting TGF-β superfamily (e.g. sotatercept)
* Prior participation in another interventional clinical study with medicinal products within 30 days or 5 half-lives prior to Screening, whichever is longer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in PVR (Pulmonary Vascular Resistance) | Baseline and Week 24
  Evaluate the effect of KER-012 on pulmonary hemodynamics compared to Placebo in participants on background pulmonary arterial hypertension (PAH) therapy

SECONDARY OUTCOMES:
Change from Baseline in the 6MWD | Through week 24 (primary treatment period) and Through week 96 (extension period)
  Evaluate the effect of KER-012 on exercise capacity compared to Placebo in participants on background PAH therapy
Incidence of treatment-emergent adverse events (TEAEs) | Through week 24 (primary treatment period) and Through week 96 (extension period)
  A TEAE is any untoward medical occurrence in a study participant occurring after the initiation of a study treatment that does not necessarily have to have a causal relationship with this treatment. A TEAE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Number of treatment-related TEAEs | Through week 24 (primary treatment period) and Through week 96 (extension period)
  A treatment-related TEAE is any untoward medical occurrence in a study participant occurring after the initiation of a study treatment that has a causal relationship with this treatment.
Number of discontinuations due to TEAEs | Through week 24 (primary treatment period) and Through week 96 (extension period)
  A treatment-related TEAE is any untoward medical occurrence in a study participant occurring after the initiation of a study treatment that has a causal relationship with this treatment. A TEAE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Change from baseline in Systolic and Diastolic Blood Pressure | Through week 24 (primary treatment period) and Through week 96 (extension period)
  Systolic and Diastolic blood pressure measured in mmHg
Change from baseline in QTcF intervals | Through week 24 (primary treatment period) and Through week 96 (extension period)
  QTcF intervals measured in msec via ECGs
Incidence of Antidrug Antibodies (ADA) | Through week 24 (primary treatment period) and Through week 96 (extension period)
  The amount of ADA measured in serum
Evaluate the changes from baseline in the concentration of the PAH biomarker, NT-proBNP in blood samples | Up to week 24 (primary treatment period) and up to Week 96 (extension period)
  Change from Baseline in NT-proBNP by visit
Evaluate the effect of KER-012 on pulmonary hemodynamics compared to Placebo in participants on background PAH therapy- mPAP | Up to week 24 (primary treatment period) and up to Week 96 (extension period)
  Change from Baseline in mean pulmonary artery pressure (mPAP)
Evaluate the effect of KER-012 on pulmonary hemodynamics compared to Placebo in participants on background PAH therapy- CO | Up to week 24 (primary treatment period) and up to Week 96 (extension period)
  Change from Baseline in cardiac output (CO)
Evaluate the effect of KER-012 on pulmonary hemodynamics compared to Placebo in participants on background PAH therapy- PAWP | Up to week 24 (primary treatment period) and up to Week 96 (extension period)
  Change from Baseline in pulmonary artery wedge pressure (PAWP)
Evaluate improvement in functional assessment of KER-012 compared to Placebo in participants on background PAH therapy | Up to week 24 (primary treatment period) and up to Week 96 (extension period)
  Proportion of participants who achieved improvement from Baseline in NYHA FC/WHO by visit
Number of participants who experienced events indicative of clinical worsening of pulmonary arterial hypertension (PAH) | Up to week 24 (primary treatment period) and up to Week 96 (extension period)
  Events that indicate clinical worsening of PAH include death, non-elective PAH-related hospitalization and/or right heart failure inclusive of lung or heart/lung transplant, or atrial septostomy, need to initiate an approved PAH SOC rescue therapy, or functional deterioration (worsened WHO Functional Class AND 15% decrease in 6MWD).
Population PK predicted maximum concentration (Cmax) of KER-012 | Through week 24 (primary treatment period) and Through week 96 (extension period)
  Cmax is a measure of the maximum concentration of a drug in the serum after the dose is given.
Population PK predicted Area under concentration curve (AUC) of KER-012 | Through week 24 (primary treatment period) and Through week 96 (extension period)
  AUC is a measure of the area under the serum concentration curve after dose is given.
Evaluate improvement in risk stratifications of KER-012 in participants on background PAH therapy | Up to week 24 (primary treatment period) and up to Week 96 (extension period)
  Proportion of participants who achieve improvement/or maintain low risk in ESC/ ERC 4-strata risk category assessment

CONTACTS AND LOCATIONS:
Locations (55):
- United States (16):
  - TROPOS Study Site 111, Scottsdale, Arizona
  - TROPOS Study Site 107, Tucson, Arizona
  - Site PI TROPOS Study Site 104, Stanford, California
  - TROPOS Study Site 105, Torrance, California
  - TROPOS Study Site 108, Jacksonville, Florida
  - TROPOS Study Site 100, Kansas City, Kansas
  - TROPOS Study Site 110, Louisville, Kentucky
  - TROPOS Study Site 103, Boston, Massachusetts
  - TROPOS Study Site 109, Boston, Massachusetts
  - TROPOS Study Site 101, Ann Arbor, Michigan
  - TROPOS Study Site 115, St Louis, Missouri
  - TROPOS Study Site 114, Albuquerque, New Mexico
  - TROPOS Study Site 113, Cincinnati, Ohio
  - TROPOS Study Site 106, Charleston, South Carolina
  - TROPOS Study Site 112, Dallas, Texas
  - TROPOS Study Site 102, Houston, Texas
- Australia (6):
  - TROPOS Study Site 805, Melbourne, Victoria
  - TROPOS Study Site 807, Auchenflower
  - TROPOS Study Site 804, Camperdown
  - TROPOS Study Site 800, Darlinghurst
  - TROPOS Study Site 803, New Lambton Heights
  - TROPOS Study Site 801, Sydney
- Brazil (3):
  - TROPOS Study Site 200, Blumenau
  - TROPOS Study Site 202, Porto Alegre
  - TROPOS Study Site 201, São Paulo
- TROPOS Study Site 320, Le Kremlin-Bicêtre, France
- Germany (6):
  - TROPOS Study Site 341, Giesen
  - TROPOS Study Site 340, Hanover
  - TROPOS Study Site 343, Heidelberg
  - TROPOS Study Site 344, Homburg
  - TROPOS Study Site 342, Leipzig
  - TROPOS Study Site 345, Regensburg
- Poland (6):
  - TROPOS Study Site 704, Gdansk
  - TROPOS Study Site 701, Krakow
  - TROPOS Study Site 705, Lodz
  - TROPOS Study Site 702, Otwock
  - TROPOS Study Site 703, Poznan
  - TROPOS Study Site 706, Poznan
- Portugal (4):
  - TROPOS Study Site 403, Almada
  - TROPOS Study Site 402, Coimbra
  - TROPOS Study Site 400, Lisbon
  - TROPOS Study Site 401, Porto
- South Korea (4):
  - TROPOS Study Site 881, Incheon
  - TROPOS Study Site 883, Seoul
  - TROPOS Study Site 882, Seoul
  - TROPOS Study Site 880, Seoul
- Spain (4):
  - TROPOS Study Site 412, Barcelona
  - TROPOS Study Site 413, Barcelona
  - TROPOS Study Site 410, Madrid
  - TROPOS Study Site 411, Santander
- Taiwan (2):
  - TROPOS Study Site 891, Kaohsiung City
  - TROPOS Study Site 890, Taipei
- United Kingdom (3):
  - TROPOS Study Site 441, Glasgow
  - TROPOS Study Site 442, London
  - TROPOS Study Site 440, London

IPD SHARING:
Plan to Share IPD: Undecided